CLINICAL TRIAL: NCT06511193
Title: Chronicling the COPD Patient Journey and Change in Impact of a Single Inhaler Combination Therapy on COPD Symptoms, Quality of Life and Exacerbations Following Initiation of Budenoside/Glycopyrronium/Formoterol [BGF](CHRONICLES COPD)
Brief Title: Chronicling the COPD Patient Journey and Change in COPD Symptoms, Quality of Life and Exacerbations Following Initiation of Budenoside/Glycopyrronium/Formoterol [BGF]
Acronym: CHRONICLES
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Asthma Research Group Inc. (Unknown); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: D5980R00105
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD;; readmissions;; maintenance therapy;; triple therapy;; real-world evidence;; mortality;; cardiopulmonary events,; exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Budenoside/Glycopyrronium/Formoterol: Patients with COPD who initiate BGF as prescribed by physician per the approved country-specific label and reimbursement criteria
  Interventions: Drug: Budenoside/Glycopyrronium/Formoterol

INTERVENTIONS:
Drug: Budenoside/Glycopyrronium/Formoterol — Patients with COPD who initiate BGF as prescribed by physician per the approved country-specific label and reimbursement criteria

SUMMARY:
The CHRONICLES study will investigate the change in clinical and patient reported outcomes after six-months of treatment with Budenoside/Glycopyrronium/Formoterol [BGF] in a real-world setting.

DETAILED DESCRIPTION:
This is a prospective, open label, non-interventional, single network of clinical practice centers study that will be conducted in routine clinical care in the pulmonary/ primary care practitioner (PCP) care setting in Ontario, Canada. Eligible patients will be enrolled into the study only following the treating physician's decision and patient agreement to initiate treatment with BGF. Patients will be observed for up to 6 months post-treatment initiation with BGF.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of COPD
* COPD patients in the Best Care Network who have a CAT score >=10
* Age >=35 at time of enrolment
* Minimum 12-month recorded prior medical history for patients
* Physician decision and patient agreement to initiate treatment with Breztri based on routine care (and in accordance with label and reimbursement criteria)
* Ability to read English and to provide consent to inclusion in the study

Exclusion Criteria:

* Diagnosis of asthma
* Dementia or other health issues related to memory
* Inability to use inhalers
* COPD due to documented α-1 antitrypsin deficiency
* Previous treatment with triple fixed-dose combination therapy in 12 months prior to screening visit
* Hospitalisation due to COPD exacerbation within the last 30 days prior to enrolment
* Pregnancy or lactation period
* Participation in an ongoing clinical interventional or observational trial for another COPD medication (or completed another trial within last 30 days of initiating BGF)
* Patient self-reporting or a physician record with an active COVID-19 infection at time of enrolment or hospitalized due to COVID-19 infection in the last 60 days
* Previous enrolment in this study

Ages: 35 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe COPD who are eligible for BGF therapy may be enrolled by physicians in primary care setting. The decision to start treatment with BGF must be made by the treating physician according to the subjects' medical need and a positive benefit/risk balance. The decision to prescribe BGF must be independent of enrolment into the study, is determined by the treating physician and should be taken according to the standard of current best medical practice and national guidelines.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in the COPD Assessment Test (CAT) score | 12 weeks after treatment initiation
  To estimate the change in COPD health status in patients initiating BGF after 12 weeks

SECONDARY OUTCOMES:
Demographic and clinical characteristics at baseline | At baseline
  To describe the demographic and clinical characteristics of patients in the study
Change from baseline in CAT score after 24 weeks of treatment | 24 weeks from treatment initiation
  To estimate the change in COPD health status after 24 weeks from treatment initiation
Change in patient quality of life as measured by EQ-5D-5L at 12 and 24 weeks post-treatment initiation | 12 and 24 weeks after treatment initiation
  To estimate the change in patient quality of life after 12 and 24 weeks of treatment initiation
Change in measures of sleep quality using CASIS (COPD and Asthma Sleep Impact Scale) at weeks 12 and 24 | 12 and 24 weeks of treatment initiation
  To estimate change in sleep quality following introduction of BGF
Percent responders of the CAT [MID=2] after 12 weeks treatment compared to baseline | 12 weeks treatment compared to baseline
  To describe the Responder Rate based on the CAT after 12 weeks of initiating treatment with BGF
The annualized rate of moderate and severe exacerbations that occurred within the previous year is collected at the baseline visit and the number of moderate and severe exacerbations occurring during the study is collected at the final visit | Baseline (12 months prior to initiating BGF) and during the follow-up period (up to 6 months))
  To describe and compare the rate of moderate and severe exacerbations

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/